CLINICAL TRIAL: NCT05816863
Title: Clinical Study of Pabolizumab for Neoadjuvant Immunotherapy of Locally Advanced Microsatellite-unstable Gastric Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Zhaode Bu, Zhaode Bu. MD, Peking University Cancer Hospital & Institute
Other Study IDs: LGH2021374
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Gastric Cancer; Gastric Adenocarcinoma
Keywords: PD-1; immuno-oncology; pabolizumab; neoadjuvant; immunotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental: pabolizumab
  Interventions: Drug: pabolizumab

INTERVENTIONS:
Drug: pabolizumab — pabolizumab IV every 3 weeks (q3w)

SUMMARY:
Our study is aim to evaluate the efficacy and safety of pabolizumab in neoadjuvant immunotherapy of locally advanced microsatellite-unstable gastric adenocarcinoma.

DETAILED DESCRIPTION:
Patients with microsatellite-unstable gastric adenocarcinoma cannot benefit from chemotherapy, According to the guideline of the Chinese Society of Clinical Oncology, It is not recommended to receive chemotherapy for patients with microsatellite-unstable gastric cancer, therefore, immunotherapy is the only hope for those patients.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG 0-1.
2. Gastroscopy confirmed adenocarcinoma of the gastroesophageal junction or stomach and biopsy pathology confirmed adenocarcinoma of the stomach.
3. Advanced gastric cancer as assessed by ultrasonography and/or gastric CT (cT3-T4b, Nany, M0).
4. Biopsy tissues with IHC indicates deficient mismatch repair(dMMR),that is, the loss of at least one of the four proteins ,MSH1, MSH2, MSH6, PMS2; or gene detection implies MSI-H;
5. Subjects must have at least one measurable lesion in accordance with RECIST v1.1. A lesion previously treated with local therapies such as radiotherapy can be considered a target lesion if there is objective evidence of progression in the lesion.
6. Is willing to provide tissue from a tumor lesion at baseline and at time of surgery.
7. Has life expectancy of greater than 6 months.
8. Adequate organ function.

Exclusion Criteria:

1. Female participants who are pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the screening visit through180 days after the last dose of chemotherapy or through 120 days after the last dose of pembrolizumab, whichever is greater.
2. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
3. as a known additional malignancy that is progressing or has required active treatment within the past 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ that have undergone potentially curative therapy are not excluded.
4. Any disease requiring systemic treatment. Local replacement steroids are permitted
5. Subjects with active, known or suspected autoimmune disease, or a medical history of autoimmune disease, with the exceptions of the following: vitiligo, alopecia, Grave disease, psoriasis or eczema not requiring systemic treatment within the last 2 years, hypothyroidism (caused by autoimmune thyroiditis) only requiring steady doses of hormone replacement therapy and type I diabetes only requiring steady doses of insulin replacement therapy, or completely relieved childhood asthma that requires no intervention in adulthood, or primary diseases that will not relapse unless triggered by external factors.
6. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
7. Known history of active tuberculosis (TB).
8. Serious infections within 4 weeks prior to the first dose of study drug, including but not limited to complications requiring hospitalization, sepsis or severe pneumonia.
9. An active infection requiring systemic therapy.
10. Subjects with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 2000 IU/ mL or active hepatitis C virus (HCV) should be excluded. Subjects with non-active HBsAg carriers, treated and stable hepatitis B (HBV DNA <500 IU/ mL) , and cured hepatitis C can be enrolled. Subjects with positive HCV antibodies are eligible only if the HCV RNA test results are negative.
11. Known history of testing positive for human immunodeficiency virus (HIV).
12. Any conditions that, in the investigator's opinion, may put subjects treated with the study drug at risks, or interfere with the evaluation of study drug or subject safety, or the interpretation of results.
13. Known history of allergy or hypersensitivity to Pabolizumab or any of its components

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced microsatellite-unstable gastric adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | Up to approximately 15 Weeks (Time of surgery)
  pCR is defined as absence of viable tumor (pT0pT0N0) in examined tissue

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 71 months.
  Overall survival is defined as the time from randomization to death due to any cause.
Progression free survival (PFS) | 3 years.
  The time from registration to the date of disease progression or death resulting from any cause.
R0 resection rate | Within 4 weeks following the operation.
  Proportion of patients who achieved R0 resection.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China